CLINICAL TRIAL: NCT05243134
Title: The Influence of Anatomic Deformities on the Clinical Efficacy in the Patients With Patellar Dislocation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2021423
Record Dates: First submitted 2021-11-23; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-09

CONDITIONS: Patellar Dislocation; Anatomic Abnormality; Trochlear Dysplasia; Femoral Anteversion; Treatment; Sport Injury
Keywords: Patellar dislocation; Anatomic deformity; trochlear dysplasia; treatment
MeSH Terms: conditions — Patellar Dislocation; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Patients with at least one type of anatomic deformity
  Interventions: Other: Collect the clinical data
- Control group: Patients without anatomic deformity
  Interventions: Other: Collect the clinical data

INTERVENTIONS:
Other: Collect the clinical data — We analyze the influence of the anatomic deformity on the clinical efficacy at the follow-up.

SUMMARY:
All the data of patients with patellar dislocation will be collected to evaluate the anatomic deformities. The data includes X-ray, CT, MRI examinations, medical records, and physical examination information. Finally, we correlate the anatomic deformities with clinical efficacy. To search for the risk factors that lead to patellar dislocation and influence the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

-Patients with patellar dislocation.

Exclusion Criteria:

* Patients with significant ligamentous knee injury.
* Previous fracture or surgery of the lower limb.
* Patellar dislocation caused by car accidents or other high-energy force directly on the patella.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with patellar dislocation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with redislocation of their patella after surgery as confirmed by clinical physical examination | Three years after surgery
  We can determine patellar redislocation by physical examination. In participants with redislocation of their patella, the patella (kneecap) slips out of its normal position. Often the knee is partly bent, painful and swollen.The patella is also often felt and seen out of place. We recored the number of participants with redislocation of their patella after surgery.
International Knee Documentation Committee(IKDC) score | Three years after surgery
  The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. The knee history form and surgical documentation form are provided for convenience. All researchers are required to complete the subjective knee evaluation and knee examination form. Instructions for scoring the subjective knee evaluation form and the knee examination form are provided on the back of the forms. Total score 100, ≥75 being considered excellent.
Magnatic Resonance Imaging evaluation | Three years after surgery
  All patients undergoing anterior cruciate ligament reconstruction underwent MRI imaging evaluation of both knees. Use International Cartilage Repair Society(ICRS) score to evaluate, total score is 12, classified into four grades,grade Ⅰ: normal (12), grade Ⅱ: nearly normal (8-11), grade Ⅲ: abnormal (4-7), grade Ⅳ: severely abnormal (1-3).

SECONDARY OUTCOMES:
Skeletal force line and various angles by X-ray evaluation | Preoperative
  X-ray was used to evaluate the skeletal force line and various angles of patients. Use Qvadriceps Angle to evaluate quadriceps force line and patellar ligament force line. The normal Angle is 18-22° for the adult standing position.Above or below this range is considered abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lin, Study Director — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu Z, Song Y, Deng R, Ye J, Wang X, Wang H, Yu JK. CT and MRI measurements of tibial tubercle lateralization in patients with patellar dislocation were not equivalent but could be interchangeable. Knee Surg Sports Traumatol Arthrosc. 2023 Jan;31(1):349-357. doi: 10.1007/s00167-022-07119-8. Epub 2022 Sep 11. PMID 36088618